CLINICAL TRIAL: NCT02724150
Title: Low Dose Against High Dose of Proton Pump Inhibitors in Treatment Acute Peptic Ulcer Bleeding
Brief Title: Comparison of Low Against High Regimen of Proton Pump Inhibitors for Treatment of Acute Peptic Ulcer Bleeding
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Damascus Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G2
Record Dates: First submitted 2016-03-14; First posted 2016-03-31 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Gastroduodenal Ulcer; Marginal Ulcer; Peptic Ulcer Hemorrhage
Keywords: Gastroduodenal Ulcer; Marginal Ulcer; Peptic Ulcer Hemorrhage; Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer; Peptic Ulcer Hemorrhage | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omeprazole High dose (Active Comparator): Omeprazole 80 mg loading dose,then 8mg/h IV continuous infusion for 3 days
  Interventions: Drug: Omeprazole High dose
- Omeprazole Low Dose (Experimental): Omeprazole 80 mg loading dose IV then 40 mg two times per day IV for 3 days
  Interventions: Drug: Omeprazole Low dose

INTERVENTIONS:
Drug: Omeprazole High dose — High regimen of Proton Pump Inhibitors in treatment of bleeding ulcer 80 mg loading dose then 8 mg/h iv for 3 days
  Arms: Omeprazole High dose
Drug: Omeprazole Low dose — low regimen of Proton Pump Inhibitors in treatment bleeding ulcer 80 mg loading dose then 40 mg two times per day for 3 days
  Arms: Omeprazole Low Dose

SUMMARY:
Evaluate the efficacy of Two different regimens of proton pump inhibitors High against Low in the management of acute peptic ulcer bleeding

DETAILED DESCRIPTION:
Evaluate the efficacy of Two different regimens of proton pump inhibitors in the management of acute peptic ulcer bleeding First: loading dose 80 mg then 8mg/h iv continuous infusion for 3 days Second Loading dose 80 mg the 40 mg every 12 h for 3 days

ELIGIBILITY:
Inclusion Criteria:

* High risk ulcers defined according to the Forrest classification With respect to high-risk stigmata,
* active bleeding was defined as a continuous blood spurting (Forrest IA)
* oozing (Forrest IB) from the ulcer base.
* A non-bleeding visible vessel at endoscopy was defined as a discrete protuberance at the ulcer base(Forrest IIA).
* An adherent clot was one that was resistant to forceful irrigation or suction (Forrest IIB).

Exclusion Criteria:

* ulcer was malignant
* non ulcerative bleeding such as angiodysplasia , a Mallory-Weiss tear....

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 month

SECONDARY OUTCOMES:
Rebleeding | one month
  recurrent melena (black, tarry stool) or recurrent Hematemesis or coffee-ground emesis or recurrent hematochezia after begin treatment
Surgery | one month
  need for surgery
Length of hospital stay | one month
Blood transfusions | one month
  number of transfusion blood unites during admission

CONTACTS AND LOCATIONS:
Overall Officials: Marouf Alhalabi, MD, Principal Investigator — Damascus Hospital
Locations (1):
- Damascus Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Undecided